CLINICAL TRIAL: NCT06440330
Title: Define Predictors for Posttransplant Diabetes Mellitus Study
Acronym: DECODE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); University Ghent (Other); Universitaire Ziekenhuizen KU Leuven (Other); HUB (Unknown); Université Catholique de Louvain (Other); Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Sponsor
Other Study IDs: 5469
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Post-transplant Diabetes Mellitus; Kidney Transplant; Complications
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: continuous glucose monitoring — continuous glucose monitoring will be used during the first 14 days post-transplantation

SUMMARY:
The primary aim of this prospective, multicentre study is to develop an accurate and convenient tool to predict the risk of PTDM at 3 months post-transplant, based on information on the day of transplantation (day 0).

In order to create such model, we will start by identifying individual predictor variables at the day of transplantation and subsequently explore the optimal combination of these predictors in multivariable models.

Secondary objectives include:

* Compare the performance of the model based on predictor variables at day 0 with existing models for prediction of PTDM (Chakkera, San Antonio Diabetes Prediction Model and Framingham Offspring Study Diabetes Mellitus algorithm)
* Explore the glucose level evolution during the first 2 weeks after transplantation using continuous glucose monitoring, and its relationship with baseline patient characteristics and immunosuppressant drug use.
* Evaluate the added value of incorporating information on glucose levels in the first and second weeks post-transplant to improve the PTDM prediction model.
* Identify predictors for early post-transplant hyperglycemia (first 2 weeks post-transplantation)
* Explore the correlation between early post-transplant hyperglycemia (fasting glycemia, pre-dinner glycemia) and PTDM at 3 months

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with end stage kidney disease undergoing kidney transplantation with a deceased or living donor
* Signed informed consent
* Initial therapy with at least tacrolimus and corticosteroids

Exclusion Criteria:

* Patients with a diagnosis of diabetes mellitus (either type 1 or type 2) prior to kidney transplantation
* Treatment with GLP1-RA for weight losing purposes
* Patients receiving a multi-organ transplantation
* ABO incompatibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients without known pre-existing diabetes.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-transplant diabetes mellitus | at 10-13 weeks post-transplantation
  Post-transplant diabetes mellitus diagnosis based on the need for glucose lowering therapy or 2h-OGTT value of >=200mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- UZA, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No